CLINICAL TRIAL: NCT01543477
Title: POST-AUTHORISATION SAFETY COHORT OBSERVATION OF RETACRIT (EPOETIN ZETA) ADMINISTERED SUBCUTANEOUSLY FOR THE TREATMENT OF RENAL ANAEMIA (PASCO II)
Brief Title: Post-Authorisation Safety Cohort Observation of RetacritTM (Epoetin Zeta) Administered Subcutaneously for the Treatment of Renal Anaemia
Acronym: PASCO II
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: EPOE-09-11; C1111006 (Other: Alias Study Number); PASCO II (Other: Alias Study Number)
Record Dates: First submitted 2012-02-21; First posted 2012-03-05 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Renal Anemia; Pregnancy; Lactation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pre-dose serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group

SUMMARY:
The purpose of this study is to estimate the incidence of Pure Red Cell Aplasia (PRCA), neutralising antibodies, lack of efficacy, and thromboembolic events under treatment with Retacrit™ (epoetin zeta) administered subcutaneously in patients with renal anaemia. The other key objective of this study is to obtain information on adverse drug reactions (ADR) associated with Retacrit™ (epoetin zeta), use of epoetin zeta during pregnancy and lactation and data on long term use.

DETAILED DESCRIPTION:
This is a non-interventional, multi-centre, longitudinal observation with a defined population using a prospective cohort design to estimate the incidence of Pure Red Cell Aplasia (PRCA), neutralising antibodies, lack of efficacy, and thromboembolic events under treatment with Retacrit™ (epoetin zeta) administered subcutaneously in patients with renal anaemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently under treatment with Retacrit™ (epoetin zeta) administered subcutaneously for renal anaemia.
* Informed consent given in writing after being provided with detailed information about the characteristics of this observation by the physician.
* Patients expected to be available for 3 years of observation

Exclusion Criteria:

* Any contraindications as per the current Summary of Product Characteristics (SPC) of Retacrit™

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients currently under treatment with Retacrit (epoetin zeta) administered subcutaneously for renal anaemia.
Sampling Method: Non-Probability Sample
Enrollment: 4501 (Actual)
Dates: Start 2010-07-07 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Incidence Rate of Adverse Events of Special Interest | 156 weeks
  Ongoing routine doctor visits for 156 weeks

SECONDARY OUTCOMES:
Adverse drug reactions | 156 weeks
  Descriptive evaluation including incidence rates of adverse drug reactions.
Information on treatment with Retacrit during pregnancy and lactation | 156 weeks
Data on long term use | 156 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (176):
- Bulgaria (14):
  - MHAT "Dr. Tota Venkova"AD, Gabrovo
  - MHAT "Dr. Stamen Iliev"AD, Montana
  - UMHAT "Georgi Stranski" EAD, Pleven
  - Dutchmed Dialysis Clinic (in the building of 5 DCC), Plovdiv
  - MHAT Plodiv AD, Plovdiv
  - MHAT "Dr. Bratan Shukerov" AD, Smolyan
  - Fifth MHAT EAD, Sofia
  - Acibadem City Clinic Tokuda Hospital EAD MHAT "Tokuda Hospital Sofia", Sofia
  - University Hospital Lozenets, Sofia
  - UMHAT "Alexandrovska" EAD, Sofia
  - SHATPD "Prof. Ivan Mitev"EAD, Sofia
  - DCC "Sveta Anna" Sofia, Sofia
  - Kidney center - Medical center EOOD, Varna
  - UMHAT "Sveta Marina"EAD, Varna
- Croatia (9):
  - County Hospital Cakovec, Čakovec
  - General Hospital Dubrovnik, Dubrovnik
  - General Hospital Karlovac, Karlovac
  - Health Center Labin, Labin
  - University Hospital Centre Osijek, Osijek
  - General Hospital Sibenik, Šibenik
  - Health Center Umag, Umag
  - University Hospital Centre Zagreb, Zagreb
  - University Hospital Merkur, Zagreb
- Department of Renal Medicine Medicinerhuset 3 sal Aalborg University Hospital, Aalborg, Denmark
- Finland (3):
  - Div. of Nephrology, Helsinki University HospitalHUS Kirurginen sairaala, Helsinki
  - Pietarsaari Hospital Medical clinic, Jakobstad
  - Kainuu Hospital, Kajaani
- France (10):
  - CHU Amiens-Picardie Site Sud,, service de Nefrologie, Amiens (Salouel) Cedex 1
  - CHU Amiens-Picardie Site Sud, Amiens (Salouel) Cedex 1
  - Centre Hospitalier de Cahors, Cahors
  - Aura Auvergne Chamalières, Chamalières
  - Hospital Gabriel Montpied, Centre de Dialyse, Clermont-Ferrand
  - 35 Nephrologie Centre Medico Chirurgical de l'Europe, Le Port-Marly
  - Polyclinique de la Louvière, Service Hemodialyse Nephrologie CHSA Maubeuge, Lille
  - Aura Paris Plaisance, Paris
  - Aura Notre Dame de Bon Secours, Paris
  - Hopital de Rangueil, service de nephrologie, Toulouse
- Germany (46):
  - Nephrologische Gemeinschaftspraxis, Alsfeld
  - PHV Dialysezentrum Alsfeld, Alsfeld
  - MVZ DaVita Alzey GmbH, Alzey
  - Gemeinschaftspraxis Dr. Gööck & Dr. Anger, Arnstadt
  - MVZ Bad Bevensen, Bad Bevensen
  - Nephrologische Gemeinschaftspraxis, Bad Homburg
  - Nephrologsiche Praxis, Bad König
  - Internistische Praxis und Nephrologie, Bad Nauheim
  - Nieren-und Hochdruckzentrum, Bad Wildungen
  - Praxis F. Nierenkrankheiten/Tagesklinik, Berlin
  - Gesundheitszentrum HSH, Berlin
  - Alwall-Haus Dialysezentrum Berlin, Berlin
  - Dialyse am Kurfürstendamm, Berlin
  - Praxis Marsen, Cologne
  - Dialyse Centrum Darmstadt, Darmstadt
  - MVZ DaVita Dormagen GmbH, Dormagen
  - KfH Nierenzentrum, Essen
  - Praxis für Nephrologie, Frankenthal
  - Nierenzentrum Heppenheim, Heppenheim an der Bergstrasse
  - Praxisklinik-Dialysezentrum Herne DOKUSAN Gesellschaft für medizinische Studien mbH & Co. KG, Herne
  - DaVita Elsterland, Herzberg
  - Dialyse T. Menzer Homberg-Efze, Homberg (Efze)
  - Nephrologische Gemeinschaftspraxis und Dialysezentrum, Hoyerswerda
  - Gemeinschaftspraxis Grahl und Johnen, Hürth-Hermülheim
  - Westpfalz-Klinikum Kaiserslautern, Kaiserslautern
  - Nieren- und Hochdruckzentrum Kiel, Kiel
  - Medizinisches Versorgungszentrum MVZ Diaverum Kleve GmbH, Kleve
  - Praxis Dres. Schoenwald und Beck, Langenfeld
  - Nephrologische Praxis, Langenselbold
  - Nierenzentrum Leverkusen, Leverkusen
  - Dialysezentrum Ludwigslust, Ludwigslust
  - Nephrologische Gemeinschaftspraxis, Lübeck
  - Märkische Kliniken GmbH Klinikum Lüdenscheid, Lüdenscheid
  - Dialysezentrum Stadtfeld, Magdeburg
  - Nephrologische Praxis, Mayen
  - Nephrologisches Zentrum, Mettmann
  - Nephrologische Gemeinschaftspraxis, Mühlhausen
  - MVZ DaVita Viersen GmbH, Nettetal
  - ze:ro Dialysezentren und Gemeinschaftspraxis, Neustadt
  - Nephrologisches- und Dialysezentrum Niebüll, Niebüll
  - Klinikum Ernst von Bergmann, Potsdam
  - Dialysezentrum, Quedlinburg
  - Gemeinschaftspraxis Schuerfeld Moeller Henrich, Saarlouis
  - Städtisches Klinikum Solingen Abt. Nephrologie - Innere Medizin, Solingen
  - Dialysezentrum Tangermünde, Tangermünde
  - Deutsche Klinik fuer Diagnostik Department of Nephrology, Wiesbaden
- Greece (44):
  - General Hospital "Asklipeiio Voulas", Voula, Attica
  - General Hospital of Rhodes, Agioi Apostoloi
  - General Hospital of Agios Nikolaos, Agios Nikolaos, Crete
  - Private Physician, Agrinio
  - Office of Eleni Stefanopoulou/Private Physician, Aigáleo
  - University General Hospital of Alexandroupoli, Alexandroupoli
  - Polikliniki Athinon, Athens
  - Therapeutical Department "ATTIKO", Athens
  - General Hospital Gennimata, Athens
  - General Hospital "Alexandra", Athens
  - Errikos Ntinan Hospital, Athens
  - Kyanos Stavros, Athens
  - Aretaiion Hospital, Athens
  - General University Hospital "ATTIKO", Athens
  - General Hospital of Athens "A.Fleming", Athens
  - Private Physician, Athens
  - General Hospital of Chania, Chania, Crete
  - Didimoticho General Hospital, Didimoticho
  - Drama General Hospital, Drama
  - Edessa General Hospital, Edessa
  - General Hospital of Filiates, Filiátes
  - General Hospital of Grevena, Grevená
  - Kavala General Hospital, Kavala
  - General Hospital of Komotini Sismanogleio, Komotini
  - Private Physician, Kozani
  - General Hospital of Kyparissia, Kyparissía
  - Private Physician, Lamia
  - General University Hospital of Larisa, Larissa
  - General Clinic Eftichios Patsidis, Larissa
  - General Hospital of Mesologgi, Mesologgi
  - Private Physician, Nea Raidestos, Thessaloniki
  - General Hospital Agios Andreas, Pátrai
  - General Hospital of Prolemaida, Ptolemaida
  - Serres general Hospital, Serres
  - AHEPA University Hospital, Thessaloniki
  - Ippokrateion General Hospital, Thessaloniki
  - Private Physician, Thessaloniki
  - Papageorgiou General Hospital, Thessaloniki
  - "Diavalkaniko" Therareutical Center, Thessaloniki
  - Therapeutical Department of Thermi, Thessaloniki
  - Papanikolaou General Hospital, Thessaloniki
  - Private Physician, Véria
  - Thessaliki Nosileutiki EPE, Volos
  - Private Physician, Voula
- Merlin Park Dialysis Unit, Galway, Ireland
- Italy (33):
  - Presidio ospesdaliero G.CRISCUOLI - UO DIALISI, Sant'Angelo dei Lombardi, Avellino
  - Policlinico S. Marco di Istituti Ospedalieri Bergamaschi, U.O. Nefrologia e Dialisi, Zingonia- Osio Sotto, Bergamo
  - "Presidio Ospedaliero" di Soverato - Servizio Dialisi, Soverato Marina, Catanzaro
  - Presidio Ospedaliero S. GIUSEPPE e MELORIO AUSL CE/2 S. - U.O. Nefrologia e Dialisi, Santa Maria Capua Vetere, CE
  - Azienda Ospedaliera S. Anna, Cona-Ferrara, Ferrara
  - U.O.C. Nefrologia e Dialisi Ospedale degli Infermi-S.Miniato-USL 11 Empoli, San Miniato, PISA
  - U.O. Nefrologia e Dialisi, Azienda Ospedaliero-Universitaria Ospedali Riuniti, Ancona
  - Ospedali Riuniti Anzio-Nettuno, Nefrologia e Dialisi ASL RMH, Anzio (RM)
  - Centro Dialisi Nefrologia - Ospedale S. Donato Arezzo, Arezzo
  - Dipartimento di Nefrologia- Ospedale Mazzoni, Ascoli Piceno
  - P.O. S.G. Moscati, Aversa (NA)
  - OSPEDALE MAGGIORE DI CHIERI - ASL TO 5 - S.C. Nefrologia e Dialisi, Chieri (TO)
  - AOU Careggi Hospital Firenze, Florence
  - Ospedale della Misericordia USL9, Grosseto
  - Dipartimento di Nefrologia Ospedale Versilia-Viareggio (Lucca), Lido Di Camaiore (Lucca)
  - U.O. Nefrologia Lucca, Lucca
  - U.O. Nefrologia e Dialisi ULSS12, Mestre
  - Ospedale Niguarda Cà Granda - U.O. Nefrologia e Dialisi e Terapia Medica del Trapianto Renale, Milan
  - Universita degli Studi di Napoli Federico II - Dipartimento di Patologia Sistematica, Naples
  - A.O. MONALDI- Dept nephrology and Dialysis, Napoli
  - Azienda Ospedaliera di Rilievo Nazionale "Antonio Cardarelli" - U.O. S. C. Nefrologia ed Emodialisi, Napoli
  - Azienda Ospedaliera Universitaria della Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - ASL SA 1 P.O. Umberto I - U.O.C. di NEFROLOGIA E DIALISI, Nocera Inferiore (SA)
  - Ospedale SANTA MARIA DELLA PIETA - U.O.C. di NEFROLOGIA E DIALISI, Nola (NA)
  - Dipartimento di Medicina -DIMED- Policlinico Padova, Padua
  - Fondazione S. Maugeri - IRCCS Clinica del Lavoro e della Riabilitazione,, Pavia
  - UO Nefrologia, trapianti e dialisi SSN EDIFICIO 30A Azienda Ospedaliera Universitaria Pisa, PISA (Cisanello)
  - U.O.C. Nefrologia e Dialisi - Ospedale "Del Ceppo", Pistoia
  - U.O.C. Nefrologia e Dialisi Azienda Ospedaliera, San Sebastiano
  - U.O.C. Nefrologia, Dialisi e Trapianto - Azienda Ospedaliera Universitaria Senese, Siena
  - A.O.U. San Giovanni Battista di Torino - S.C. di Nefrologia, Dialisi e Trapianto, Torino
  - Ospedale Martini - S.C. Nefrologia E Dialisi, Torino
  - Ospedale San Giovanni Bosco - Struttura Complessa Nefrologia e Dialisi, Torino
- Spain (10):
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Xanit Hospital Internacional, Benalmádena, Málaga
  - Hospital Lluis Alcanyis, Xàtiva, Valencia
  - Fundació Puigvert, Barcelona
  - Hospital de Barcelona, Barcelona
  - Hospital Universitario de Leon, León
  - Hospital central della Cruz Roja, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Parc Taulí, Sabadell
  - Hospital Virgen de la Concha, Zamora
- Sweden (4):
  - Karlskoga Lasarett, Karlskoga
  - Linköpings Universitetssjukhus, Linköping
  - Karolinska University Hospital, Stockholm
  - Njurmedicinska kliniken, Danderyds sjukhus, Stockholm
- Kings College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.